CLINICAL TRIAL: NCT01749397
Title: A Phase I Trial of the Combination of the PARP Inhibitor ABT-888 With Intraperitoneal Floxuridine (FUDR) in Epithelial Ovarian, Primary Peritoneal and Fallopian Tube Cancers
Brief Title: Veliparib and Floxuridine in Treating Patients With Metastatic Epithelial Ovarian, Primary Peritoneal Cavity, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02767; NCI-2012-02767 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1114; 9182 (Other: Mayo Clinic in Rochester); 9182 (Other: CTEP); P30CA015083 (NIH); P50CA136393 (NIH); U01CA069912 (NIH); UM1CA186686 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: interventions — Floxuridine; 5-fluoro-2'-deoxyuridine; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (veliparib and floxuridine) (Experimental): Patients receive veliparib PO BID on days 1-10 and floxuridine IP on days 3-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Floxuridine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Veliparib

INTERVENTIONS:
Drug: Floxuridine — Given IP
  Other Names: 2''-Deoxy-5-fluorouridine; 5-Fluoro-2''-deoxyuridine; 5-Fluorodeoxyuridine; 5-Fluorouracil deoxyriboside; 5-FUdR; FDUR; Floxuridin; Fluorodeoxyuridine; Fluorouridine Deoxyribose; Fluoruridine Deoxyribose; FUdR; WR-138720
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Veliparib — Given IV
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given together with floxuridine in treating patients with epithelial ovarian, primary peritoneal cavity, or fallopian tube cancer that has spread to other places in the body. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as floxuridine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving veliparib together with floxuridine may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of the combination of ABT-888 (veliparib) and intraperitoneal (IP) floxuridine in adult patients with advanced ovarian, primary peritoneal or fallopian tube cancer.

SECONDARY OBJECTIVES:

I. To describe the adverse event profile associated with this treatment combination.

II. To assess for preliminary evidence of efficacy, such as tumor responses, of the treatment combination.

III. To assess progression free survival (PFS) in the maximum tolerated dose (MTD) cohort.

TERTIARY OBJECTIVES:

I. Assess the pharmacokinetic profile of ABT-888 and floxuridine when given in combination.

II. Assess whether the presence of mutations in the homologous recombination pathway or loss of expression of non-homologous end joining (NHEJ) components correlates with response to floxuridine + ABT-888.

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive veliparib orally (PO) twice daily (BID) on days 1-10 and floxuridine IP on days 3-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian, primary peritoneal or fallopian tube malignancy that is metastatic and for which standard curative measures do not exist
* Disease confined to the intraperitoneal and retroperitoneal cavity; Note: nodal disease below the diaphragm, implants adherent to the surface of the liver or intrahepatic lesions will not be exclusionary; patients remain eligible if all intrahepatic tumor is debulked or ablated by the time treatment is initiated
* EXPANSION PHASE ONLY: Evaluable or measurable disease with the largest nodule measuring less than 5 cm in greatest dimension by radiographic imaging after debulking procedure
* Candidate for and willingness to have a surgically placed intraperitoneal catheter and tissue acquisition at the time of port placement; note: if an intraperitoneal catheter is already in place, a tumor biopsy will still be required; a guided core-needle biopsy is sufficient in these cases
* Able to swallow and absorb the medication
* Obtained =< 7 days prior to registration: Absolute neutrophil count (ANC) >= 1500/mm^3
* Obtained =< 7 days prior to registration: Platelets (PLT) >= 100,000/mm^3
* Obtained =< 7 days prior to registration: Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Obtained =< 7 days prior to registration: Creatinine =< 1.5 x institutional ULN
* Obtained =< 7 days prior to registration: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 3 x institutional ULN
* Obtained =< 7 days prior to registration: Hemoglobin (Hgb) > 9.0 mg/dl
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Ability to provide informed written consent
* Life expectancy >= 12 weeks
* Women of childbearing potential only: negative pregnancy test done =< 7 days prior to registration

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy; note: patients with recurrent platinum-sensitive ovarian, primary peritoneal or fallopian tube will be allowed, if the investigator believes the study treatment is a better alternative to initiation platinum-based chemotherapy, such as patients with a prior platinum allergy or low volume disease for whom platinum-based therapy is deferred until a later date
* More than 4 prior chemotherapy regimens; note: repeat use of regimens count as 1 prior regimen; switching front-line therapy regimens (for example, from intraperitoneal to intravenous therapy) for reasons other than progression will count as 1 prior therapy; bevacizumab and other 'targeted' agents will count in the total number of prior regimens; vaccine therapies will not count in the total of prior therapies
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 28 days prior to registration
  * Mitomycin C/nitrosoureas =< 42 days prior to registration
  * Immunotherapy =< 28 days prior to registration
  * Biologic therapy =< 28 days prior to registration
  * Radiation therapy =< 28 days prior to registration
  * Investigational therapy or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA] approved indication and in the context of a research investigation) =< 28 days prior to registration
  * Prior poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor therapy
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* Significant cardiovascular disease defined as congestive heart failure (New York Heart Association class III or IV cardiac disease), angina pectoris requiring nitrate therapy or recent myocardial infarction (=< 6 months prior to registration)
* Metastatic disease outside the intraperitoneal cavity and retroperitoneum, intrahepatic lesions, or pleural effusions; significant ascites precluding catheter placement; exception: intrahepatic lesions removed or planning to be removed during the debulking procedure
* Any of the following:

  * Nursing women
  * Pregnant women
  * Women of childbearing potential who are unwilling to employ adequate contraception (non-barrier method)
* Immunocompromised patients (other than that related to the use of corticosteroids) with the exception of patients known to be human immunodeficiency virus (HIV) positive and have a cluster of differentiation 4 (CD4) count > 400 and do not require antiretroviral therapy
* Receiving any other investigational agent that would be considered a treatment for the primary neoplasm
* Other active malignancy =< 1 year prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2017-10-20 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 21 days
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion. This will provide an indication of the level of tolerance for this treatment combination in this patient group.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 months
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion. This will provide an indication of the level of tolerance for this treatment combination in this patient group.
Incidence of toxicities assessed using CTCAE version 4.0 | Up to 3 months
  Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Incidence of non-hematologic toxicities evaluated via the CTC standard toxicity grading | Up to 3 months
  Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Incidence of hematologic toxicity | Up to 3 months
  Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Response profile assessed using Response Evaluation Criteria in Solid Tumors | Up to 3 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Time until any treatment related toxicity | Up to 3 months
  Will be summarized descriptively.
Time until treatment related grade 3+ toxicity | Up to 3 months
  Will be summarized descriptively.
Time until hematologic nadirs (white blood cell, absolute neutrophil count [ANC], platelets) | Up to 3 months
  Will be summarized descriptively.
Time to progression | Up to 3 months
  Will be summarized descriptively.
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months
  Will be summarized descriptively.

OTHER OUTCOMES:
Pharmacokinetic parameters | Prior to administration of floxuridine and veliparib, 0.25, 0.5, 1, 2, 4, 6, and 9 hours (day 1 and 3 of course 1), prior to administration of floxuridine and veliparib on days 4-5 of course 1, and prior to administration of veliparib on day 6 course 1
  Data will be presented in mean and standard deviation in table form.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea E Wahner Hendrickson, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Washington University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri